CLINICAL TRIAL: NCT04255719
Title: Unilateral Pallidal vs Unilateral Subthalamic Nucleus Deep Brain Stimulation in the Same Patient With Parkinson Disease: A Randomized Controlled Trial
Brief Title: Unilateral GPi vs Unilateral STN DBS in the Same Patient With PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, chief physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020 UPS study
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease; Deep Brain Stimulation; Globus Pallidus Interna; Subthalamic Nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Throughout the study, all participants, independent raters/evaluators and statisticians will be blind to the treatment conditions and parameter configurations. Independent raters who are blind to the conditions will be responsible for the conduct of all the assessments. Participants are blind to the treatment conditions. Movement disorders clinician responsible for programming are blind to the study protocol. They are simply told to adjust parameter to optimize therapeutic effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral DBS of the subthalamic nucleus (STN) (Experimental): To deliver unilateral STN DBS, bilateral stimulation will be turned off for three hours, and then turn on the unilateral STN DBS. The STN stimulation will be programmed as previous parameter configuration with optimal therapeutic benefits. Participants will be asked to complete a comprehensive set of assessments under unilateral STN stimulation in the off-medication state. 45 minutes after taking regular medication, participants need to complete the second set of assessments in the on-medication state.
  Interventions: Procedure: DBS
- Unilateral DBS of the globus pallidus interna (GPi) (Experimental): To deliver unilateral GPi DBS, bilateral stimulation will be turned off for three hours, and then turn on the unilateral GPi DBS. The study protocol is identical to the intervention of unilateral STN DBS but it was done on a different day.
  Interventions: Procedure: DBS

INTERVENTIONS:
Procedure: DBS — Unilateral DBS for treatment of patients with PD

SUMMARY:
The subthalamic nucleus (STN) and globus pallidus interna (GPi) are two main targets in the deep brain stimulation (DBS) treatment for Parkinson's disease (PD). Large randomized controlled trials, in which patients of comparable clinical and demographics were randomized to either GPi DBS or STN DBS, have demonstrated equal effects of both targets in motor symptom improvement, the superiority of STN DBS in the medication reduction and the potential advantage of GPi DBS for cognitive, psychiatric and axial aspects. Unfortunately, in such a highly heterogeneous disease of PD, many of these randomized controlled trials didn't include sufficient subjects and thereby yielded inconsistent results. Moreover, most studies are investigating the difference between GPi and STN in different patients.

In order to address the problem, an intra-patient comparison will be made by investigating the acute turning-on effects of unilateral STN stimulation versus unilateral GPi stimulation on axial symptoms, cognition and also cardinal symptoms within each individual patient who received the treatment of combined unilateral STN and contralateral GPi DBS. Axial symptoms including gait, balance and posture, motor symptoms and cognition are comprehensively assessed under two treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease
* Aged between 55 and 75 years, both male and female
* Patients who have undergone combined unilateral STN and contralateral GPi DBS for more than 6 months
* A Hoehn-Yahr (H-Y) stage of less than 4 in the off-medication state
* A left-extremity to right-extremity ratio of less than 0.15 on the Unified Parkinson's Disease Rating Scale part Ⅲ (UPDRS-Ⅲ) in the both off-medication and on-medication states

Exclusion Criteria:

* History of serious psychosis
* History of intractable epilepsy (i.e., seizures)
* Diagnosed by the investigators that patients with severe cardiac, liver and kidney diseases, or other serious health conditions
* Dementia (A Mini-Mental State Examination (MMSE) score of < 24), inability to comprehend the experimental protocol or voluntarily provide informed consent
* Lack of cooperation
* Additional reasons for exclusion at the discretion of the clinical investigator
* Poorly controlled depression or anxiety
* Past history of suicidal attempt

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Difference in Timed Up-and-Go (TUG) task scores between treatment conditions in the on- and off- medication states | 6 months
  Timed Up-and-Go task is a well-defined objective gait measurement. The task requires an individual to stand up, walk 5 m, turn, walk back, and sit down. The time taken to complete the test is strongly correlated with the level of functional mobility. This test will be videotaped and scored by two blinded neurologists.

SECONDARY OUTCOMES:
Differences in total Uniﬁed Parkinson's Disease Rating Scale Part Ⅲ (UPDRS Ⅲ) scores between two treatment conditions in the on- and off- medication states | 6 months
  Uniﬁed Parkinson's Disease Rating Scale Part Ⅲ measures the motor severity of Parkinson's disease. UPDRS Ⅲ score has a range of 0 (no symptoms) to 132 (severe disease symptoms).
Differences in Burg Balance Scale (BBS) scores between two treatment conditions in the on- and off- medication states. | 6 months
  Burg Balance Scale measures patients' static and dynamic balance abilities. BBS score has a range of 0 (severe balance problems) to 56 (no balance problems).
Differences in postural angles between two treatment conditions in the on- and off- medication states. | 6 months
  The measurement of postural angles is the same as the paper (Yamada et al) published in J Neurol Neurosurg Psychiatry
Differences in Water Swallow Test (WST) scores between treatment conditions in the on- and off- medication states. | 6 months
  The Water Swallow Test is frequently used in clinical practice as a functional assessment to detect dysphagia, with stage 1 indicating severe dysphagia and stage 6 indicating normal swallowing function.
Differences in Swallowing Disturbance Questionnaire (SDQ) scores between treatment conditions in the on- and off- medication states. | 6 months
  The Swallowing Disturbance Questionnaire is created as a self-rated dysphagia screening tool in PD, with a range of 0 (normal swallowing function) to 42 (severe dysphagia).
Differences in voice parameters between treatment conditions in the on- and off- medication states. | 6 months
  Voice recording at a sampling rate of 44.1 kHz using 16-bit quantification will be conducted in a sound-treated room using a microphone and a digital voice recorder with a mouth-to-microphone distance of 15 cm. The recorded voices will then be used for a composit acoustic analysis.
Differences in Voice Handicap Index (VHI) between treatment conditions in the on- and off- medication states. | 6 months
  The Voice Handicap Index is a self-administered instrument, comprising 30 items on voice-related dysfunction. VHI has a range of 0 (normal voice function) to 120 (severe voice dysfunction).

CONTACTS AND LOCATIONS:
Locations (1):
- Functional neurosurgery of Shanghai jiaotong university affiliated Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamada K, Shinojima N, Hamasaki T, Kuratsu J. Subthalamic nucleus stimulation improves Parkinson's disease-associated camptocormia in parallel to its preoperative levodopa responsiveness. J Neurol Neurosurg Psychiatry. 2016 Jul;87(7):703-9. doi: 10.1136/jnnp-2015-310926. Epub 2015 Sep 30. PMID 26424897
- [Background] Lizarraga KJ, Luca CC, De Salles A, Gorgulho A, Lang AE, Fasano A. Asymmetric neuromodulation of motor circuits in Parkinson's disease: The role of subthalamic deep brain stimulation. Surg Neurol Int. 2017 Oct 24;8:261. doi: 10.4103/sni.sni_292_17. eCollection 2017. PMID 29184712